CLINICAL TRIAL: NCT02285114
Title: A Phase 2/3, Open-Label, Multi-Cohort Switch Study to Evaluate Emtricitabine/Tenofovir Alafenamide (F/TAF) in HIV-1 Infected Children and Adolescents Virologically Suppressed on a 2-NRTI-Containing Regimen
Brief Title: Study To Evaluate Emtricitabine/Tenofovir Alafenamide (F/TAF) in Human Immunodeficiency Virus 1 (HIV-1) Infected Children and Adolescents Virologically Suppressed on a 2-Nucleoside/Nucleotide Reverse Transcriptase Inhibitor (2-NRTI)-Containing Regimen
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-311-1269; 2015-001339-19 (EudraCT Number)
Record Dates: First submitted 2014-11-04; First posted 2014-11-06 (Estimated); Results first posted 2021-01-12 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: HIV-1
Keywords: emtricitabine; FTC; tenofovir; TDF; antiretroviral; adolescents; children; pediatric; TAF

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- F/TAF+3rd ARV Agent (Cohort 1) (Experimental): Participants between 12 to < 18 years of age and ≥ 35 kg in body weight will switch their current 2-NRTI containing regimen to F/TAF (200/25 mg for unboosted 3rd agent and 200/10 mg for boosted 3rd agent) while continuing on their 3rd ARV agent for 48 weeks.
  Interventions: Drug: F/TAF; Drug: 3rd ARV agent
- F/TAF+3rd ARV Agent (Cohort 2, Part A - Group 1) (Experimental): Participants between 6 to < 12 years of age and ≥ 25 kg in body weight must be on a boosted protease inhibitor (PI) as their 3rd ARV agent and will switch their current 2-NRTI regimen to F/TAF 200/25 mg while continuing on their boosted PI for 48 weeks.
  Interventions: Drug: F/TAF; Drug: Boosted PIs
- F/TAF+3rd ARV Agent (Cohort 2, Part A - Group 2) (Experimental): Participants between 2 to < 12 years of age and between 17 kg to < 25 kg in body weight must be on a boosted protocol specified 3rd ARV agent and will switch their current 2-NRTI containing regimen to F/TAF 120/15 mg while continuing their 3rd ARV agent for 48 weeks.
  Interventions: Drug: F/TAF; Drug: 3rd ARV agent
- FTC/TAF+3rd ARV Agent (Cohort 3, Part A) (Experimental): Participants between 2 to < 6 years of age will receive F/TAF plus a 3rd ARV agent through 48 weeks.
  Interventions: Drug: F/TAF; Drug: 3rd ARV agent
- FTC/TAF+3rd ARV Agent (Cohort 4, Part A) (Experimental): Participants between 1 month to < 2 years of age will receive F/TAF plus a 3rd ARV agent through 48 weeks.
  Interventions: Drug: F/TAF; Drug: 3rd ARV agent
- F/TAF+3rd ARV Agent (Cohort 2, Part B - Group 1) (Experimental): Screening will be initiated for Part B following confirmation of TAF dose in Part A. Approximately 10 additional total participants will be enrolled across all Part B cohorts and will receive F/TAF while continuing their 3rd ARV agent through 48 weeks.
  Interventions: Drug: F/TAF; Drug: 3rd ARV agent
- F/TAF+3rd ARV Agent (Cohort 2, Part B - Group 2) (Experimental): Screening will be initiated for Part B following confirmation of TAF dose in Part A. Approximately 10 additional total participants will be enrolled across all Part B cohorts and will receive F/TAF while continuing their 3rd ARV agent through 48 weeks.
  Interventions: Drug: F/TAF; Drug: 3rd ARV agent
- FTC/TAF+3rd ARV Agent (Cohort 3, Part B) (Experimental): Screening will be initiated for Part B following confirmation of TAF dose in Part A. Approximately 10 additional total participants will be enrolled across all Part B cohorts and will receive F/TAF while continuing their 3rd ARV agent through 48 weeks.
  Interventions: Drug: F/TAF; Drug: 3rd ARV agent
- FTC/TAF+3rd ARV Agent (Cohort 4, Part B) (Experimental): Screening will be initiated for Part B following confirmation of TAF dose in Part A. Approximately 10 additional total participants will be enrolled across all Part B cohorts and will receive F/TAF while continuing their 3rd ARV agent through 48 weeks.
  Interventions: Drug: F/TAF; Drug: 3rd ARV agent
- FTC/TAF+3rd ARV Agent (Extension Phase) (Experimental): After completion of 48 weeks, all participants will be given the option to participate in an extension phase of the study. Gilead will provide F/TAF until a) the participant turns 18 and F/TAF is commercially available for use in adults in the country in which the participant is enrolled or, b) F/TAF becomes commercially available for pediatric use in the country in which the participant is enrolled or, c) Gilead Sciences elects to terminate development of F/TAF in the applicable country.
  Interventions: Drug: F/TAF; Drug: 3rd ARV agent

INTERVENTIONS:
Drug: F/TAF — F/TAF tablets administered orally once daily
Drug: 3rd ARV agent — A 3rd antiretroviral (ARV) agent may include one of the following: allowed boosted 3rd ARV agents: lopinavir (LPV), atazanavir (ATV), darunavir (DRV); Allowed unboosted 3rd ARV agents: efavirenz (EFV), raltegravir (RAL), dolutegravir (DTG), or nevirapine (NVP)
  Arms: F/TAF+3rd ARV Agent (Cohort 1); F/TAF+3rd ARV Agent (Cohort 2, Part A - Group 2); F/TAF+3rd ARV Agent (Cohort 2, Part B - Group 1); F/TAF+3rd ARV Agent (Cohort 2, Part B - Group 2); FTC/TAF+3rd ARV Agent (Cohort 3, Part A); FTC/TAF+3rd ARV Agent (Cohort 3, Part B); FTC/TAF+3rd ARV Agent (Cohort 4, Part A); FTC/TAF+3rd ARV Agent (Cohort 4, Part B); FTC/TAF+3rd ARV Agent (Extension Phase)
Drug: Boosted PIs — Allowed boosted PIs: LPV, ATV, DRV.
  Arms: F/TAF+3rd ARV Agent (Cohort 2, Part A - Group 1)

SUMMARY:
The primary objective of this study is to confirm the TAF dose and to evaluate the pharmacokinetics (PK) of TAF, safety, and tolerability of F/TAF in children and adolescents with HIV-1 who are virologically suppressed (defined as having < 50 copies/mL of HIV-1 ribonucleic acid (RNA) for a period of at least 6 months) while on a stable 2 NRTI containing regimen.

DETAILED DESCRIPTION:
A minimum of 100 participants in total (across all cohorts) aged 1 month to <18 years of age will be enrolled to receive F/TAF. The study will proceed in sequential cohorts as follows: Cohort 1 will switch their current 2-NRTI-containing regimen to F/TAF while continuing on their 3rd ARV agent through 48 weeks; Cohorts 2, 3, and 4 must be on a boosted protease inhibitor (PI) (Cohort 2 only) or any other 3rd ARV agent and will switch their current 2-NRTI-containing regimen to F/TAF while continuing their boosted PI or 3rd ARV agent through 48 weeks. A minimum of 10 participants each in Groups 1 and 2 of Cohort 2, and Cohorts 3 and 4, who are on boosted-ATV as their 3rd ARV agent will be enrolled. Cohorts 2, 3, and 4 will be enrolled by cohort into a two-part study (Parts A and B).

After completion of 48 weeks, all participants will be given the option to participate in an extension phase of the study. Gilead will provide F/TAF until a) The participant turns 18 years old and F/TAF is commercially available for use in adults in the country in which the participant is enrolled or b), F/TAF becomes commercially available for pediatric use in the country in which the participant is enrolled or c), Gilead Sciences elects to terminate development of F/TAF in the applicable country.

However, Cohort 2 (Part B), Cohorts 3 and 4 were not conducted as planned.

ELIGIBILITY:
Key Inclusion Criteria:

* Human immunodeficiency virus 1 (HIV-1) infected male and female adolescents and children aged 1 month to < 18 years at baseline/Day 1 (according to requirements of the enrolling cohort)
* Must be able to give written assent prior to any screening evaluations
* Parent or guardian able to give written informed consent prior to any screening evaluations and willing to comply with study requirements
* Body weight at screening as follows:

  * Cohort 1: ≥ 35 kg
  * Cohort 2, Group 1: ≥ 25 kg
  * Cohort 2, Group 2: 17 kg to < 25 kg
  * Cohort 3: to be updated per a protocol amendment
  * Cohort 4: to be updated per a protocol amendment
* Currently on a stable 2-nucleoside/nucleotide reverse transcriptase inhibitor (NRTI) containing regimen that includes a 3rd antiretroviral (ARV) agent for ≥ 6 consecutive months prior to screening
* Plasma HIV-1 ribonucleic acid (RNA) levels < 50 copies/mL for ≥ 6 consecutive months preceding the screening visit
* No opportunistic infection within 30 days of study entry (at baseline/Day 1)
* A negative serum β-human chorionic gonadotropin (HCG) pregnancy test is required for females of childbearing potential only

Key Exclusion Criteria:

* An acquired immunodeficiency syndrome (AIDS) - indicator condition with onset within 30 days prior to screening
* Life expectancy of < 2 years
* Active, serious infections (other than HIV-1 infection) requiring parenteral antibiotic or antifungal therapy within 30 days prior to baseline/Day 1
* Evidence of active pulmonary or extra-pulmonary tuberculosis disease within 3 months of the screening visit
* Active hepatitis C virus (HCV) infection defined as positive for HCV antibody and having detectable HCV RNA
* Positive hepatitis B surface antigen or other evidence of active hepatitis B virus (HBV) infection.
* Have any serious or active medical or psychiatric illness which, in the opinion of the Investigator, would interfere with treatment, assessment, or compliance with the protocol.
* Pregnant or lactating females
* Have history of significant drug sensitivity or drug allergy
* Have previously participated in an investigational trial involving administration of any investigational agent, other than TDF, within 30 days prior to the study dosing

NOTE: Other protocol defined Inclusion/ Exclusion criteria may apply.

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2015-01-20 (Actual); Primary Completion 2019-11-04 (Actual); Study Completion 2024-12-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (8):
- United States (4):
  - University of California Los Angeles, Los Angeles, California
  - Children's Hospital Colorado, Aurora, Colorado
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Seattle Children's Hospital, Seattle, Washington
- Hospital del Nino, Panama City, Panama
- South Africa (3):
  - Rahima Moosa Mother and Child Hospital, Johannesburg, Coronationville
  - KIDCRU, Ward J8, Tygerberg Children's Hospital, Cape Town
  - Be Part Yoluntu Centre, Cape Town

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at https://www.gileadclinicaltrials.com/transparency-policy#Commitment
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: https://www.gileadclinicaltrials.com/transparency-policy#Commitment

REFERENCES:
- [Background] Chen JS, Saez-Llorens X, Castano E, Patel F, Melvin A, McFarland EJ, et al. Safety, Pharmacokinetics, and Efficacy of FTC/TAF in HIV-Infected Adolescents (12-18 years) [Poster 843]. Conference on Retroviruses and Opportunistic Infections (CROI); 2018 04-07 March; Boston, MA.
- [Background] Castano E, Deville J, Zuidewind P, Vedder J, German P, Mathias A, et al. PK and Safety of F/TAF With Boosted 3rd Agents in Children With HIV [Abstract 54]. International Workshop on HIV & Pediatrics 2020; 2020 November 16-17 Virtual.
- [Background] Cox S, Porter D, White K, Graham H, Pikora C, Callebaut C. Tenofovir Alafenamide-Based Regimens: A Pooled Resistance Analysis in Pediatric Participants [Abstract 4]. International Workshop on HIV Pediatrics 2019; 2019 July 19-20; San Francisco, CA.
- [Background] Rakhmanina N, Cunningham C, Cotton M, Natukunda E, Rodriguez C, Gaur A, et al. Weight Trajectory in Children and Adolescents Who Switched to TAF-Based Regimens [Abstract 56]. International Workshop on HIV & Pediatrics 2020; 2020 November 16-17; Virtual.
- [Background] Sharma S, Gupta S, Majeed SR, Strehlau R, Hellstrom E, Liu Y, et al. Exposure-Safety of Tenofovir in Pediatric HIV Infected Participants: Comparison of Tenofovir Alafenamide and Tenofovir Disoproxil Fumarate [Abstract 23]. Presented at International Workshop on HIV Pediatrics 2018; 2018 July 20-21; Amsterdam, The Netherlands.
- [Background] Cotton M, Cunningham C, Natukunda E, Rodriguez C, Gaur A, Kosalaraksa P, et al. Lack of Influence of Pubertal Stage on Safety and TFV Pharmacokinetics in TAF-based Regimens [Abstract 43]. International Workshop on HIV Pediatrics 2019; 2019 July 19-20; San Francisco, CA.
- [Background] Andreatta K, Cox S, Chokephaibulkit K, Rodriguez C, Liberty A, Natukunda E, et al. Preexisting and Post-Baseline Resistance Analyses in Pooled Pediatric Studies of Emtricitabine/Tenofovir Alafenamide (F/TAF)-Based Antiretroviral Therapy. 12th IAS Conference on HIV Science; 2023 23-26 July; Brisbane, Australia.
- [Background] Rakhmanina N, Gaur A, Deville JG, Kosalaraksa P, Strehlau R, Natukunda E, et al. Bone Mineral Density in Children With HIV 1 Receiving TAF Based Antiretroviral Therapy [Abstract 948]. Conference on Retroviruses and Opportunistic Infections (CROI); 2024 03-06 March; Denver, CO.
- [Background] Mujuru H, Strehlau R, Kosalaraksa A, Deville JG, Pan M, Vieira VA, et al. Week 24 Outcomes of F/TAF Plus Cobicistat-Boosted Protease Inhibitors in Children ≥ 2 Years and ≥ 14 kg [Abstract] Presented at Conference on Retroviruses an Opportunistic Infections (CROI); 2025 09-12 March, San Francisco, CA.
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=GS-US-311-1269

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 49 participants were screened. Participants were enrolled at study sites in Panama, South Africa, and United States.
Pre-assignment Details: No participant was enrolled in Cohort 2 (Part B: Groups 1 and 2), and Cohorts 3 and 4 (Parts A and B). Data is reported only for Cohorts 1 and 2 (Part A: Groups 1 and 2). The study had a main treatment phase of 48 weeks and extension phase.
  It was prespecified to analyze Cohort 1 together as both treatments (F/TAF 200/10 mg with boosted 3rd ARV and F/TAF 200/25 mg with unboosted 3rd ARV) were expected to have a similar effect on efficacy and safety for target population.
Groups:
- Main Phase: F/TAF+3rd ARV Agent (Cohort 1): Participants between 12 to < 18 years of age and ≥ 35 kg body weight received emtricitabine/tenofovir alafenamide (F/TAF) 200/10 mg fixed-dose combination (FDC) tablet (with boosted 3rd antiretroviral (ARV) agent) or F/TAF 200/25 mg FDC tablet (with unboosted 3rd ARV agent) orally once daily for 48 weeks. Allowed boosted 3rd ARV agents: lopinavir (LPV), atazanavir (ATV), darunavir (DRV); Allowed unboosted 3rd ARV agents: efavirenz (EFV), raltegravir (RAL), dolutegravir (DTG), or nevirapine (NVP).
- Main Phase: F/TAF+3rd ARV Agent (Cohort 2, Part A - Group 1): Participants between 6 to < 12 years of age and ≥ 25 kg body weight received F/TAF 200/25 mg FDC tablet orally once daily while continuing on their boosted protease inhibitor (PI) for 48 weeks. Allowed boosted PIs: ATV, LPV or DRV.
- Main Phase: F/TAF+3rd ARV Agent (Cohort 2, Part A - Group 2): Participants between 2 to < 12 years of age and 17 to < 25 kg body weight received F/TAF 120/15 mg FDC orally once daily while continuing on their 3rd ARV agent for 48 weeks. Allowed boosted 3rd ARV agents: LPV, ATV, DRV; Allowed unboosted 3rd ARV agents: EFV, RAL, DTG, or NVP.
- Extension Phase: F/TAF+3rd ARV Agent (Cohort 1): After completion of 48 weeks, all participants were given the option to participate in an extension phase of the study to continue with F/TAF+3rd ARV Agent. Gilead provided F/TAF until a) the participant turned 18 and F/TAF was commercially available for use in adults in the country in which the participant was enrolled or, b) F/TAF became commercially available for pediatric use in the country in which the participant was enrolled or, c) Gilead Sciences elected to terminate development of F/TAF in the applicable country. The maximum exposure was 438.9 weeks. Allowed boosted 3rd ARV agents: LPV, ATV, DRV. Allowed unboosted 3rd ARV agents: EFV, RAL, DTG, or NVP.
- Extension Phase: F/TAF+3rd ARV Agent (Cohort 2, Part A - Group 1): After completion of 48 weeks, all participants were given the option to participate in an extension phase of the study to continue with F/TAF+3rd ARV agent. Gilead provided F/TAF until a) the participant turned 18 and F/TAF was commercially available for use in adults in the country in which the participant was enrolled or, b) F/TAF became commercially available for pediatric use in the country in which the participant is enrolled or, c) Gilead Sciences elected to terminate development of F/TAF in the applicable country. The maximum exposure was 315.0 weeks. Allowed boosted PIs: ATV, LPV or DRV
- Extension Phase: F/TAF+3rd ARV Agent (Cohort 2, Part A -Group 2): After completion of 48 weeks, all participants were given the option to participate in an extension phase of the study to continue with F/TAF+3rd ARV Agent. Gilead provided F/TAF until a) the participant turned 18 and F/TAF was commercially available for use in adults in the country in which the participant was enrolled or, b) F/TAF became commercially available for pediatric use in the country in which the participant was enrolled or, c) Gilead Sciences elected to terminate development of F/TAF in the applicable country. The maximum exposure was 103.1 weeks. Allowed boosted 3rd ARV agents: LPV, ATV, DRV; Allowed unboosted 3rd ARV agents: EFV, RAL, DTG, or NVP.
Period: Main Phase
Arm/Group | Main Phase: F/TAF+3rd ARV Agent (Cohort 1) | Main Phase: F/TAF+3rd ARV Agent (Cohort 2, Part A - Group 1) | Main Phase: F/TAF+3rd ARV Agent (Cohort 2, Part A - Group 2) | Extension Phase: F/TAF+3rd ARV Agent (Cohort 1) | Extension Phase: F/TAF+3rd ARV Agent (Cohort 2, Part A - Group 1) | Extension Phase: F/TAF+3rd ARV Agent (Cohort 2, Part A -Group 2)
Started | 29 | 9 | 3 | 0 | 0 | 0
Completed | 28 | 7 | 2 | 0 | 0 | 0
Not Completed | 1 | 2 | 1 | 0 | 0 | 0
Not completed — Investigator's Discretion | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Enrolled but Never Treated | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrew Consent | 0 | 0 | 1 | 0 | 0 | 0
Period: Extension Phase
Arm/Group | Main Phase: F/TAF+3rd ARV Agent (Cohort 1) | Main Phase: F/TAF+3rd ARV Agent (Cohort 2, Part A - Group 1) | Main Phase: F/TAF+3rd ARV Agent (Cohort 2, Part A - Group 2) | Extension Phase: F/TAF+3rd ARV Agent (Cohort 1) | Extension Phase: F/TAF+3rd ARV Agent (Cohort 2, Part A - Group 1) | Extension Phase: F/TAF+3rd ARV Agent (Cohort 2, Part A -Group 2)
Started | 0 | 0 | 0 | 28 | 7 | 2
Completed | 0 | 0 | 0 | 10 | 5 | 2
Not Completed | 0 | 0 | 0 | 18 | 2 | 0
Not completed — Investigator's Discretion | 0 | 0 | 0 | 14 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Non-compliance with Study Drug | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all participants who were enrolled in the study and had received at least one dose of study medication.
  It was prespecified to analyze data from Cohort 1 together because both treatments (F/TAF 200/10 mg with boosted 3rd ARV and F/TAF 200/25 mg with unboosted 3rd ARV) were expected to have a similar effect on the efficacy and safety for the target population.
Groups:
- F/TAF+3rd ARV Agent (Cohort 1): Participants between 12 to < 18 years of age and ≥ 35 kg body weight received emtricitabine/tenofovir alafenamide (F/TAF) 200/10 mg fixed-dose combination (FDC) tablet (with boosted 3rd antiretroviral [ARV] agent) or F/TAF 200/25 mg FDC tablet (with unboosted 3rd ARV agent) orally once daily for 48 weeks. After completion of 48 weeks, all participants were given the option to participate in the extension phase of the study to continue with F/TAF+3rd ARV agent. Gilead provided F/TAF until a) the participant turned 18 and F/TAF was commercially available for use in adults in the country in which the participant was enrolled or, b) F/TAF became commercially available for pediatric use in the country in which the participant was enrolled or, c) Gilead Sciences elected to terminate development of F/TAF in the applicable country. (Allowed boosted 3rd ARV agents: lopinavir [LPV], atazanavir [ATV], darunavir [DRV]; Allowed unboosted 3rd ARV agents: efavirenz [EFV], raltegravir [RAL], dolutegravir [DTG], or nevirapine [NVP]). The participants received the study drug up to a maximum of 438.9 weeks.
- F/TAF+3rd ARV Agent (Cohort 2, Part A - Group 1): Participants between 6 to < 12 years of age and ≥ 25 kg body weight received F/TAF 200/25 mg FDC tablet orally once daily while continuing on their boosted protease inhibitor (PI) for 48 weeks. After completion of 48 weeks, all participants were given the option to participate in the extension phase of the study to continue with F/TAF+3rd ARV agent. Gilead provided F/TAF until a) the participant turned 18 and F/TAF was commercially available for use in adults in the country in which the participant was enrolled or, b) F/TAF became commercially available for pediatric use in the country in which the participant was enrolled or, c) Gilead Sciences elected to terminate development of F/TAF in the applicable country. (Allowed boosted PIs: ATV, LPV or DRV). The participants received the study drug up to a maximum of 315.0 weeks.
- F/TAF+3rd ARV Agent (Cohort 2, Part A - Group 2): Participants between 2 to < 12 years of age and 17 to < 25 kg body weight received F/TAF 120/15 mg FDC orally once daily while continuing on their 3rd ARV agent for 48 weeks. After completion of 48 weeks, all participants were given the option to participate in the extension phase of the study to continue with F/TAF+3rd ARV agent. Gilead provided F/TAF until a) the participant turned 18 and F/TAF was commercially available for use in adults in the country in which the participant was enrolled or, b) F/TAF became commercially available for pediatric use in the country in which the participant was enrolled or, c) Gilead Sciences elected to terminate development of F/TAF in the applicable country. (Allowed boosted 3rd ARV agents: LPV, ATV, DRV; Allowed unboosted 3rd ARV agents: EFV, RAL, DTG, or NVP). The participants received the study drug up to a maximum of 103.1 weeks.
- Total: Total of all reporting groups
Arm/Group | F/TAF+3rd ARV Agent (Cohort 1) | F/TAF+3rd ARV Agent (Cohort 2, Part A - Group 1) | F/TAF+3rd ARV Agent (Cohort 2, Part A - Group 2) | Total
Number analyzed (Participants) | 28 | 9 | 3 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 14 (1.6) | 10 (1.0) | 7 (1.2) | 13 (2.6)
Age, Customized [Count of Participants; unit: Participants]
  6 to < 12 years | 0 | 9 | 3 | 12
  12 to < 15 years | 19 | 0 | 0 | 19
  15 to < 18 years | 9 | 0 | 0 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 5 | 2 | 19
  Male | 16 | 4 | 1 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 5 | 1 | 20
  Not Hispanic or Latino | 14 | 4 | 2 | 20
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 1 | 0 | 0 | 1
  Race: Black | 12 | 4 | 2 | 18
  Race: White | 3 | 0 | 0 | 3
  Race: Other | 12 | 5 | 1 | 18
Region of Enrollment [Number; unit: participants]
  Panama | 12 | 6 | 1 | 19
  South Africa | 10 | 0 | 2 | 12
  United States | 6 | 3 | 0 | 9
Human Immunodeficiency Virus, Type 1 Ribonucleic Acid (HIV-1 RNA) [Count of Participants; unit: Participants]
  < 50 copies/mL | 27 | 9 | 3 | 39
  ≥ 50 copies/mL | 1 | 0 | 0 | 1
Cluster of Differentiation 4 (CD4) Cell Count [Mean (Standard Deviation); unit: cells/µL] | 909 (242.7) | 871 (364.8) | 1209 (306.3) | 923 (282.8)
CD4 Percentage (%) [Mean (Standard Deviation); unit: percentage of lymphocytes] | 36.1 (6.40) | 36.7 (4.35) | 36.1 (3.35) | 36.2 (5.73)

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetic (PK) Parameter (Cohort 1): AUCtau of Tenofovir Alafenamide (TAF)
Description: AUCtau is defined as the area under the drug concentration versus time curve over the dosing interval.
Time Frame: Any time at Week 2 visit
Population: Participants in the Intensive PK (IPK) Analysis Set (participants who were enrolled in Cohort 1 for IPK evaluation, had received at least one dose of study medication, and had at least 1 non-missing PK concentration data for any analyte of interest (e.g., emtricitabine (FTC), TAF, and tenofovir (TFV))) with available data were analyzed.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Groups:
- F/TAF 200/10 mg+3rd ARV Agent (Cohort 1): Participants between 12 to < 18 years of age and ≥ 35 kg body weight received F/TAF 200/10 mg FDC tablet (with boosted 3rd ARV agent) orally once daily for 48 weeks. After completion of 48 weeks, all participants were given the option to participate in an extension phase of the study to continue with F/TAF+3rd ARV agent. Gilead provided F/TAF until a) the participant turned 18 and F/TAF was commercially available for use in adults in the country in which the participant was enrolled or, b) F/TAF became commercially available for pediatric use in the country in which the participant was enrolled or, c) Gilead Sciences elected to terminate development of F/TAF in the applicable country. (Allowed boosted 3rd ARV agents: LPV, ATV, DRV). The participants received the study drug up to a maximum of 438.9 weeks.
- F/TAF 200/25 mg+3rd ARV Agent (Cohort 1): Participants between 12 to < 18 years of age and ≥ 35 kg body weight received F/TAF 200/25 mg FDC tablet (with unboosted 3rd ARV agent) orally once daily for 48 weeks. After completion of 48 weeks, all participants were given the option to participate in an extension phase of the study to continue with F/TAF+3rd ARV agent. Gilead provided F/TAF until a) the participant turned 18 and F/TAF was commercially available for use in adults in the country in which the participant was enrolled or, b) F/TAF became commercially available for pediatric use in the country in which the participant was enrolled or, c) Gilead Sciences elected to terminate development of F/TAF in the applicable country. (Allowed unboosted 3rd ARV agents: EFV, RAL, DTG, or NVP). The participants received the study drug up to a maximum of 438.9 weeks.
Arm/Group | F/TAF 200/10 mg+3rd ARV Agent (Cohort 1) | F/TAF 200/25 mg+3rd ARV Agent (Cohort 1)
Number analyzed (Participants) | 9 | 9
h*ng/mL | 139.9 (113.23) | 200.6 (83.80)

2. Primary Outcome: PK Parameter (Cohort 2: Part A - Groups 1 and 2): AUCtau of TAF
Description: AUCtau is defined as the area under the drug concentration versus time curve over the dosing interval.
Time Frame: Any time at Week 2 or Week 4 visit, or within 7 days after the completion of Week 2 or Week 4 visits
Population: The IPK Analysis Set included all participants who were enrolled into the study, had received at least one dose of study medication, and had at least 1 non-missing PK concentration data for any analyte of interest (e.g., FTC, TAF, and TFV).
Measure: Mean (Standard Deviation); unit: h*ng/mL
Groups:
- F/TAF+3rd ARV Agent (Cohort 2, Part A - Group 1): Participants between 6 to < 12 years of age and ≥ 25 kg body weight received F/TAF 200/25 mg FDC tablet orally once daily while continuing on their boosted PI for 48 weeks. After completion of 48 weeks, all participants were given the option to participate in an extension phase of the study to continue with F/TAF+3rd ARV agent. Gilead provided F/TAF until a) the participant turned 18 and F/TAF was commercially available for use in adults in the country in which the participant was enrolled or, b) F/TAF became commercially available for pediatric use in the country in which the participant was enrolled or, c) Gilead Sciences elected to terminate development of F/TAF in the applicable country. (Allowed boosted PIs: ATV, LPV or DRV). The participants received the study drug up to a maximum of 315.0 weeks.
- F/TAF+3rd ARV Agent (Cohort 2, Part A - Group 2): Participants between 2 to < 12 years of age and 17 to < 25 kg body weight received F/TAF 120/15 mg FDC orally once daily while continuing on their 3rd ARV agent for 48 weeks. After completion of 48 weeks, all participants were given the option to participate in an extension phase of the study to continue with F/TAF+3rd ARV agent. Gilead provided F/TAF until a) the participant turned 18 and F/TAF was commercially available for use in adults in the country in which the participant was enrolled or, b) F/TAF became commercially available for pediatric use in the country in which the participant was enrolled or, c) Gilead Sciences elected to terminate development of F/TAF in the applicable country. (Allowed boosted 3rd ARV agents: LPV, ATV, DRV; Allowed unboosted 3rd ARV agents: EFV, RAL, DTG, or NVP). The participants received the study drug up to a maximum of 103.1 weeks.
Arm/Group | F/TAF+3rd ARV Agent (Cohort 2, Part A - Group 1) | F/TAF+3rd ARV Agent (Cohort 2, Part A - Group 2)
Number analyzed (Participants) | 9 | 3
h*ng/mL | 210.8 (97.35) | 220.2 (187.96)

3. Primary Outcome: Percentage of Participants Experiencing Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) Through Week 24
Description: An AE is any untoward medical occurrence in a clinical study participant which does not necessarily have a causal relationship with the treatment. An AE can therefore be any unfavorable and/or unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. The TEAEs were defined as any AEs with an onset date of on or after the study drug start date and no later than 30 days after permanent discontinuation of study drug or any AEs leading to premature discontinuation of study drug.
Time Frame: Baseline through Week 24
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Groups:
- F/TAF+3rd ARV Agent (Cohort 2, Part A - Group 1): Participants between 6 to < 12 years of age and ≥ 25 kg body weight received F/TAF 200/25 mg FDC tablet orally once daily while continuing on their boosted PI for 48 weeks. After completion of 48 weeks, all participants were given the option to participate in the extension phase of the study to continue with F/TAF+3rd ARV agent. Gilead provided F/TAF until a) the participant turned 18 and F/TAF was commercially available for use in adults in the country in which the participant was enrolled or, b) F/TAF became commercially available for pediatric use in the country in which the participant was enrolled or, c) Gilead Sciences elected to terminate development of F/TAF in the applicable country. (Allowed boosted PIs: ATV, LPV or DRV). The participants received the study drug up to a maximum of 315.0 weeks.
Arm/Group | F/TAF+3rd ARV Agent (Cohort 1) | F/TAF+3rd ARV Agent (Cohort 2, Part A - Group 1) | F/TAF+3rd ARV Agent (Cohort 2, Part A - Group 2)
Number analyzed (Participants) | 28 | 9 | 3
percentage of participants
  Any AEs | 82.1 | 66.7 | 66.7
  SAEs | 7.1 | 0 | 0

4. Secondary Outcome: PK Parameter (Cohort 1): Cmax of TAF, FTC, and TFV
Description: Cmax is defined as the maximum concentration of drug.
Time Frame: Any time at Week 2 visit
Population: Participants in the IPK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- F/TAF 200/10 mg+3rd ARV Agent (Cohort 1): Participants between 12 to < 18 years of age and ≥ 35 kg body weight received F/TAF 200/10 mg FDC tablet (with boosted 3rd ARV agent) orally once daily for 48 weeks. After completion of 48 weeks, all participants given the option to participate in an extension phase of the study to continue with F/TAF+3rd ARV agent. Gilead provided F/TAF until a) the participant turned 18 and F/TAF was commercially available for use in adults in the country in which the participant was enrolled or, b) F/TAF became commercially available for pediatric use in the country in which the participant was enrolled or, c) Gilead Sciences elected to terminate development of F/TAF in the applicable country. (Allowed boosted 3rd ARV agents: LPV, ATV, DRV). The participants received the study drug up to a maximum of 438.9 weeks.
Arm/Group | F/TAF 200/10 mg+3rd ARV Agent (Cohort 1) | F/TAF 200/25 mg+3rd ARV Agent (Cohort 1)
Number analyzed (Participants) | 13 | 11
ng/mL
  Cmax of TAF | 89.1 (77.63) | 139.3 (76.17)
  Cmax of FTC | 2259.2 (470.75) | 2320.0 (482.18)
  Cmax of TFV | 21.2 (4.89) | 11.6 (2.74)

5. Secondary Outcome: PK Parameter (Cohort 2: Part A - Groups 1 and 2): Cmax of TAF, FTC, and TFV
Description: Cmax is defined as the maximum concentration of drug.
Time Frame: Any time at Week 2 or Week 4 visit, or within 7 days after the completion of Week 2 or Week 4 visits
Population: Participants in the IPK Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | F/TAF+3rd ARV Agent (Cohort 2, Part A - Group 1) | F/TAF+3rd ARV Agent (Cohort 2, Part A - Group 2)
Number analyzed (Participants) | 9 | 3
ng/mL
  Cmax of TAF | 230.4 (264.70) | 232.0 (253.59)
  Cmax of FTC | 2074.4 (565.91) | 2020.0 (1151.91)
  Cmax of TFV | 55.8 (19.20) | 48.1 (8.07)

6. Secondary Outcome: PK Parameter (Cohort 1): Clast of TAF
Description: Clast is defined as the last observable concentration of drug.
Time Frame: Any time at Week 2 visit
Population: Participants in the IPK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | F/TAF 200/10 mg+3rd ARV Agent (Cohort 1) | F/TAF 200/25 mg+3rd ARV Agent (Cohort 1)
Number analyzed (Participants) | 13 | 11
ng/mL | 2.2 (0.98) | 5.5 (3.76)

7. Secondary Outcome: PK Parameter (Cohort 2: Part A - Groups 1 and 2): Clast of TAF
Description: Clast is defined as the last observable concentration of drug.
Time Frame: Any time at Week 2 or Week 4 visit, or within 7 days after the completion of Week 2 or Week 4 visits
Population: Participants in the IPK Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | F/TAF+3rd ARV Agent (Cohort 2, Part A - Group 1) | F/TAF+3rd ARV Agent (Cohort 2, Part A - Group 2)
Number analyzed (Participants) | 9 | 3
ng/mL | 2.9 (2.32) | 2.1 (0.86)

8. Secondary Outcome: PK Parameter (Cohort 1): CL/F of TAF
Description: CL/F is defined as the apparent clearance following oral administration of the drug.
Time Frame: Any time at Week 2 visit
Population: Participants in the IPK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | F/TAF 200/10 mg+3rd ARV Agent (Cohort 1) | F/TAF 200/25 mg+3rd ARV Agent (Cohort 1)
Number analyzed (Participants) | 9 | 9
L/hr | 129.8 (101.67) | 143.4 (53.55)

9. Secondary Outcome: PK Parameter (Cohort 2: Part A - Groups 1 and 2): CL/F of TAF
Description: CL/F is defined as the apparent clearance following oral administration of the drug.
Time Frame: Any time at Week 2 or Week 4 visit, or within 7 days after the completion of Week 2 or Week 4 visits
Population: Participants in the IPK Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | F/TAF+3rd ARV Agent (Cohort 2, Part A - Group 1) | F/TAF+3rd ARV Agent (Cohort 2, Part A - Group 2)
Number analyzed (Participants) | 9 | 3
L/hr | 174.3 (156.75) | 102.1 (60.75)

10. Secondary Outcome: PK Parameter (Cohort 1): Vz/F of TAF
Description: Vz/F is defined as the apparent volume of distribution of the drug following oral administration.
Time Frame: Any time at Week 2 visit
Population: Participants in the IPK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: liters
Groups:
- F/TAF 200/25 mg +3rd ARV Agent (Cohort 1): Participants between 12 to < 18 years of age and ≥ 35 kg body weight received F/TAF 200/25 mg FDC tablet (with unboosted 3rd ARV agent) orally once daily for 48 weeks. After completion of 48 weeks, all participants were given the option to participate in an extension phase of the study to continue with F/TAF+3rd ARV agent. Gilead provided F/TAF until a) the participant turned 18 and F/TAF was commercially available for use in adults in the country in which the participant was enrolled or, b) F/TAF became commercially available for pediatric use in the country in which the participant was enrolled or, c) Gilead Sciences elected to terminate development of F/TAF in the applicable country. (Allowed unboosted 3rd ARV agents: EFV, RAL, DTG, or NVP). The participants received the study drug up to a maximum of 438.9 weeks.
Arm/Group | F/TAF 200/10 mg+3rd ARV Agent (Cohort 1) | F/TAF 200/25 mg +3rd ARV Agent (Cohort 1)
Number analyzed (Participants) | 9 | 9
liters | 87.3 (60.68) | 95.3 (43.47)

11. Secondary Outcome: PK Parameter (Cohort 2: Part A - Groups 1 and 2): Vz/F of TAF
Description: Vz/F is defined as the apparent volume of distribution of the drug following oral administration.
Time Frame: Any time at Week 2 or Week 4 visit, or within 7 days after the completion of Week 2 or Week 4 visits
Population: Participants in the IPK Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | F/TAF+3rd ARV Agent (Cohort 2, Part A - Group 1) | F/TAF+3rd ARV Agent (Cohort 2, Part A - Group 2)
Number analyzed (Participants) | 9 | 3
liters | 160.8 (145.57) | 63.1 (63.39)

12. Secondary Outcome: PK Parameter (Cohort 1): AUCtau of FTC and TFV
Description: AUCtau is defined as the area under the drug concentration versus time curve over the dosing interval.
Time Frame: Any time at Week 2 visit
Population: Participants in the IPK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Groups:
- F/TAF 200/10 mg+3rd ARV Agent (Cohort 1): Participants between 12 to < 18 years of age and ≥ 35 kg body weight received F/TAF 200/10 mg FDC tablet (with boosted 3rd ARV agent) orally once daily for 48 weeks. After completion of 48 weeks, all participants were given the option to participate in an extension phase of the study. Gilead provided F/TAF until a) the participant turned 18 and F/TAF was commercially available for use in adults in the country in which the participant was enrolled or, b) F/TAF became commercially available for pediatric use in the country in which the participant was enrolled or, c) Gilead Sciences elected to terminate development of F/TAF in the applicable country. (Allowed boosted 3rd ARV agents: LPV, ATV, DRV). The participants received the study drug up to a maximum of 438.9 weeks.
Arm/Group | F/TAF 200/10 mg+3rd ARV Agent (Cohort 1) | F/TAF 200/25 mg+3rd ARV Agent (Cohort 1)
Number analyzed (Participants) | 13 | 11
h*ng/mL
  AUCtau of FTC | 14769.9 (4481.23) | 14339.8 (6099.55)
  AUCtau of TFV | 415.5 (105.92) | 193.2 (46.73)

13. Secondary Outcome: PK Parameter (Cohort 2: Part A - Groups 1 and 2): AUCtau of FTC and TFV
Description: AUCtau is defined as the area under the drug concentration versus time curve over the dosing interval.
Time Frame: Any time at Week 2 or Week 4 visit, or within 7 days after the completion of Week 2 or Week 4 visits
Population: Participants in the IPK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | F/TAF+3rd ARV Agent (Cohort 2, Part A - Group 1) | F/TAF+3rd ARV Agent (Cohort 2, Part A - Group 2)
Number analyzed (Participants) | 9 | 3
h*ng/mL
  AUCtau of FTC: number analyzed (Participants) | 8 | 3
  AUCtau of FTC | 12360.8 (2928.36) | 11171.7 (2921.64)
  AUCtau of TFV | 999.4 (409.33) | 908.2 (90.62)

14. Secondary Outcome: PK Parameter (Cohort 1): Ctau of FTC and TFV
Description: Ctau is defined as the observed drug concentration at the end of the dosing interval.
Time Frame: Any time at Week 2 visit
Population: Participants in the IPK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | F/TAF 200/10 mg+3rd ARV Agent (Cohort 1) | F/TAF 200/25 mg+3rd ARV Agent (Cohort 1)
Number analyzed (Participants) | 13 | 11
ng/mL
  Ctau of FTC | 223.4 (482.59) | 301.7 (624.77)
  Ctau of TFV | 15.7 (4.11) | 6.7 (3.00)

15. Secondary Outcome: PK Parameter (Cohort 2: Part A - Groups 1 and 2): Ctau of FTC and TFV
Description: Ctau is defined as the observed drug concentration at the end of the dosing interval.
Time Frame: Any time at Week 2 or Week 4 visit, or within 7 days after the completion of Week 2 or Week 4 visits
Population: Participants in the IPK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | F/TAF+3rd ARV Agent (Cohort 2, Part A - Group 1) | F/TAF+3rd ARV Agent (Cohort 2, Part A - Group 2)
Number analyzed (Participants) | 9 | 3
ng/mL
  Ctau of FTC: number analyzed (Participants) | 8 | 3
  Ctau of FTC | 75.4 (22.71) | 75.4 (27.63)
  Ctau of TFV | 34.8 (16.39) | 30.9 (3.53)

16. Secondary Outcome: Percentage of Participants Experiencing TEAEs and SAEs Through Week 48
Description: as for outcome 3
Time Frame: Baseline through Week 48
Population: Participants in the Safety Analysis Set were analyzed. It was prespecified to analyze data from Cohort 1 together because both treatments (F/TAF 200/10 mg with boosted 3rd ARV and F/TAF 200/25 mg with unboosted 3rd ARV) were expected to have a similar effect on the efficacy and safety for the target population.
Measure: Number; unit: percentage of participants
Arm/Group | F/TAF+3rd ARV Agent (Cohort 1) | F/TAF+3rd ARV Agent (Cohort 2, Part A - Group 1) | F/TAF+3rd ARV Agent (Cohort 2, Part A - Group 2)
Number analyzed (Participants) | 28 | 9 | 3
percentage of participants
  Any AEs | 89.3 | 77.8 | 66.7
  SAEs | 7.1 | 0 | 0

17. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 24, as Defined by the United States Food and Drug Administration (US FDA)-Defined Snapshot Algorithm
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at Week 24 was analyzed using the snapshot algorithm, which defined a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 24
Population: The Full Analysis Set included all participants who were enrolled in the study and had received at least one dose of study medication. It was prespecified to analyze data from Cohort 1 together because both treatments (F/TAF 200/10 mg with boosted 3rd ARV and F/TAF 200/25 mg with unboosted 3rd ARV) were expected to have a similar effect on the efficacy and safety for the target population.
Measure: Number; unit: percentage of participants
Arm/Group | F/TAF+3rd ARV Agent (Cohort 1) | F/TAF+3rd ARV Agent (Cohort 2, Part A - Group 1) | F/TAF+3rd ARV Agent (Cohort 2, Part A - Group 2)
Number analyzed (Participants) | 28 | 9 | 3
percentage of participants | 92.9 | 100.0 | 66.7

18. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 48, as Defined by the US FDA-Defined Snapshot Algorithm
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at Week 48 was analyzed using the snapshot algorithm, which defined a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 48
Population: Participants in the Full Analysis Set were analyzed. It was prespecified to analyze data from Cohort 1 together because both treatments (F/TAF 200/10 mg with boosted 3rd ARV and F/TAF 200/25 mg with unboosted 3rd ARV) were expected to have a similar effect on the efficacy and safety for the target population.
Measure: Number; unit: percentage of participants
Arm/Group | F/TAF+3rd ARV Agent (Cohort 1) | F/TAF+3rd ARV Agent (Cohort 2, Part A - Group 1) | F/TAF+3rd ARV Agent (Cohort 2, Part A - Group 2)
Number analyzed (Participants) | 28 | 9 | 3
percentage of participants | 89.3 | 77.8 | 66.7

19. Secondary Outcome: Change From Baseline in CD4+ Cell Count at Week 24
Time Frame: Baseline, Week 24
Population: Participants in the Full Analysis Set with available data were analyzed. It was prespecified to analyze data from Cohort 1 together because both treatments (F/TAF 200/10 mg with boosted 3rd ARV and F/TAF 200/25 mg with unboosted 3rd ARV) were expected to have a similar effect on the efficacy and safety for the target population.
Measure: Mean (Standard Deviation); unit: cells/µL
Groups:
- F/TAF+3rd ARV Agent (Cohort 1): Participants between 12 to < 18 years of age and ≥ 35 kg body weight received emtricitabine/tenofovir alafenamide (F/TAF) 200/10 mg fixed-dose combination (FDC) tablet (with boosted 3rd antiretroviral [ARV] agent) or F/TAF 200/25 mg FDC tablet (with unboosted 3rd ARV agent) orally once daily for 48 weeks. After completion of 48 weeks, all participants were given the option to participate in the extension phase of the study to continue with F/TAF+3rd ARV agent. Gilead provided F/TAF until a) the participant turned 18 and F/TAF was commercially available for use in adults in the country in which the participant was enrolled or, b) F/TAF became commercially available for pediatric use in the country in which the participant was enrolled or, c) Gilead Sciences elected to terminate development of F/TAF in the applicable country. (Allowed boosted 3rd ARV agents: lopinavir [LPV], atazanavir [ATV], darunavir [DRV]; Allowed unboosted 3rd ARV agents: efavirenz [EFV], raltegravir [RAL], dolutegravir [DTG], or nevirapine [NVP])The participants received the study drug up to a maximum of 438.9 weeks.
Arm/Group | F/TAF+3rd ARV Agent (Cohort 1) | F/TAF+3rd ARV Agent (Cohort 2, Part A - Group 1) | F/TAF+3rd ARV Agent (Cohort 2, Part A - Group 2)
Number analyzed (Participants) | 28 | 8 | 2
cells/µL | -130 (272.6) | 68 (352.5) | -299 (48.8)

20. Secondary Outcome: Change From Baseline in CD4+ Cell Count at Week 48
Time Frame: Baseline, Week 48
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | F/TAF+3rd ARV Agent (Cohort 1) | F/TAF+3rd ARV Agent (Cohort 2, Part A - Group 1) | F/TAF+3rd ARV Agent (Cohort 2, Part A - Group 2)
Number analyzed (Participants) | 28 | 7 | 2
cells/µL | -105 (162.9) | 210 (406.5) | -124 (37.5)

21. Secondary Outcome: Change From Baseline in CD4 Percentage at Week 24
Time Frame: Baseline, Week 24
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: percentage of lymphocytes
Arm/Group | F/TAF+3rd ARV Agent (Cohort 1) | F/TAF+3rd ARV Agent (Cohort 2, Part A - Group 1) | F/TAF+3rd ARV Agent (Cohort 2, Part A - Group 2)
Number analyzed (Participants) | 28 | 8 | 2
percentage of lymphocytes | -0.21 (3.840) | 1.29 (2.395) | 0.60 (5.798)

22. Secondary Outcome: Change From Baseline in CD4 Percentage at Week 48
Time Frame: Baseline, Week 48
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: percentage of lymphocytes
Arm/Group | F/TAF+3rd ARV Agent (Cohort 1) | F/TAF+3rd ARV Agent (Cohort 2, Part A - Group 1) | F/TAF+3rd ARV Agent (Cohort 2, Part A - Group 2)
Number analyzed (Participants) | 28 | 7 | 2
percentage of lymphocytes | -0.20 (3.407) | 0.70 (3.520) | 3.65 (7.283)

23. Secondary Outcome: Number of Participants With Palatability of F/TAF Formulation
Description: Palatability was reported based on the pleasant product taste as 'Yes' or 'No'. Data has been reported for Participant Response (PR) and Guardian Response (GR). Participants with missing data were reported as N/A.
Time Frame: Week 2 (for Cohort 1), Week 2 and Week 4 (for Cohort 2)
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | F/TAF+3rd ARV Agent (Cohort 1) | F/TAF+3rd ARV Agent (Cohort 2, Part A - Group 1) | F/TAF+3rd ARV Agent (Cohort 2, Part A - Group 2)
Number analyzed (Participants) | 28 | 9 | 3
Participants
  Week 2: Participant Response: Was the Study Drug Palatable?: Yes | 25 | 9 | 2
  Week 2: Participant Response: Was the Study Drug Palatable?: No | 0 | 0 | 0
  Week 2: Participant Response: Was the Study Drug Palatable?: NA | 3 | 0 | 1
  Week 4: Participant Response: Was the Study Drug Palatable?: number analyzed (Participants) | 0 | 9 | 3
  Week 4: Participant Response: Was the Study Drug Palatable?: Yes |  | 9 | 3
  Week 4: Participant Response: Was the Study Drug Palatable?: No |  | 0 | 0
  Week 4: Participant Response: Was the Study Drug Palatable?: NA |  | 0 | 0
  Week 2: Guardian Response: Was the Study Drug Palatable to the Participant?: Yes | 11 | 9 | 1
  Week 2: Guardian Response: Was the Study Drug Palatable to the Participant?: No | 0 | 0 | 0
  Week 2: Guardian Response: Was the Study Drug Palatable to the Participant?: NA | 17 | 0 | 2
  Week 4: Guardian Response: Was the Study Drug Palatable to the Participant?: number analyzed (Participants) | 0 | 9 | 3
  Week 4: Guardian Response: Was the Study Drug Palatable to the Participant?: Yes |  | 9 | 1
  Week 4: Guardian Response: Was the Study Drug Palatable to the Participant?: No |  | 0 | 0
  Week 4: Guardian Response: Was the Study Drug Palatable to the Participant?: NA |  | 0 | 2
  Week 2: Guardian Response: Did the Participant Complain of the Taste of the Tablet?: Yes | 0 | 0 | 0
  Week 2: Guardian Response: Did the Participant Complain of the Taste of the Tablet?: No | 12 | 9 | 1
  Week 2: Guardian Response: Did the Participant Complain of the Taste of the Tablet?: NA | 16 | 0 | 2
  Week 4: Guardian Response: Did the Participant Complain of the Taste of the Tablet?: number analyzed (Participants) | 0 | 9 | 3
  Week 4: Guardian Response: Did the Participant Complain of the Taste of the Tablet?: Yes |  | 0 | 0
  Week 4: Guardian Response: Did the Participant Complain of the Taste of the Tablet?: No |  | 9 | 1
  Week 4: Guardian Response: Did the Participant Complain of the Taste of the Tablet?: NA |  | 0 | 2

24. Secondary Outcome: Number of Participants With Acceptability of F/TAF Formulation
Description: Acceptability has been reported for categories medication size, shape and difficulty swallowing as 'Yes' or 'No' for Participant Response (PR) and Guardian Response (GR). Participants with missing data were reported as N/A.
Time Frame: Baseline up to Week 4
Population: Participants in the Safety Analysis Set with available data were analyzed. It was prespecified to analyze data from Cohort 1 together because both treatments (F/TAF 200/10 mg with boosted 3rd ARV and F/TAF 200/25 mg with unboosted 3rd ARV) were expected to have a similar effect on the efficacy and safety for the target population.
Measure: Count of Participants; unit: Participants
Arm/Group | F/TAF+3rd ARV Agent (Cohort 1) | F/TAF+3rd ARV Agent (Cohort 2, Part A - Group 1) | F/TAF+3rd ARV Agent (Cohort 2, Part A - Group 2)
Number analyzed (Participants) | 25 | 9 | 3
Participants
  Participant Response: Was the Study Medication Size Acceptable?: Yes | 25 | 9 | 3
  Participant Response: Was the Study Medication Size Acceptable?: No | 0 | 0 | 0
  Participant Response: Was the Study Medication Size Acceptable?: N/A | 0 | 0 | 0
  Participant Response: Was the Study Medication Shape Acceptable?: Yes | 25 | 9 | 3
  Participant Response: Was the Study Medication Shape Acceptable?: No | 0 | 0 | 0
  Participant Response: Was the Study Medication Shape Acceptable?: N/A | 0 | 0 | 0
  Guardian Response: Did the Participant Have Difficulty Swallowing the Tablet?: Yes | 0 | 0 | 0
  Guardian Response: Did the Participant Have Difficulty Swallowing the Tablet?: No | 21 | 9 | 2
  Guardian Response: Did the Participant Have Difficulty Swallowing the Tablet?: N/A | 4 | 0 | 1

ADVERSE EVENTS:
Time Frame: All-cause mortality: Up to 439 weeks; Adverse events (AEs): Up to 410.4 weeks
Description: All-cause mortality: All Enrolled Analysis Set. AEs: Safety Analysis Set: all participants who had received at least 1 dose of study medication. It was prespecified to analyze data from Cohort 1 together because both treatments (F/TAF 200/10 mg+boosted 3rd ARV and F/TAF 200/25 mg+unboosted 3rd ARV) were expected to have a similar effect on efficacy and safety for target population. AEs are reported together for both phases as participants continued same medication from main to extension phase.
Groups:
- F/TAF+3rd ARV Agent (Cohort 1): Participants between 12 to < 18 years of age and ≥ 35 kg body weight received emtricitabine/tenofovir alafenamide (F/TAF) 200/10 mg fixed-dose combination (FDC) tablet (with boosted 3rd antiretroviral (ARV) agent) or F/TAF 200/25 mg FDC tablet (with unboosted 3rd ARV agent) orally once daily for 48 weeks. After completion of 48 weeks, all participants were given the option to participate in the extension phase of the study to continue with F/TAF+3rd ARV agent. Gilead provided F/TAF until a) the participant turned 18 and F/TAF was commercially available for use in adults in the country in which the participant was enrolled or, b) F/TAF became commercially available for pediatric use in the country in which the participant was enrolled or, c) Gilead Sciences elected to terminate development of F/TAF in the applicable country. (Allowed boosted 3rd ARV agents: lopinavir (LPV), atazanavir (ATV), darunavir (DRV); Allowed unboosted 3rd ARV agents: efavirenz (EFV), raltegravir (RAL), dolutegravir (DTG), or nevirapine (NVP)). The participants received the study drug up to a maximum of 438.9 weeks.
Arm/Group | F/TAF+3rd ARV Agent (Cohort 1) | F/TAF+3rd ARV Agent (Cohort 2, Part A - Group 1) | F/TAF+3rd ARV Agent (Cohort 2, Part A - Group 2)
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/9 | 0/3
Serious Adverse Events (participants affected / at risk) | 4/28 | 1/9 | 0/3
Other Adverse Events (participants affected / at risk) | 27/28 | 8/9 | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | F/TAF+3rd ARV Agent (Cohort 1) (N=28) | F/TAF+3rd ARV Agent (Cohort 2, Part A - Group 1) (N=9) | F/TAF+3rd ARV Agent (Cohort 2, Part A - Group 2) (N=3)
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0
Stab wound (Injury, poisoning and procedural complications) | 1 | 0 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | F/TAF+3rd ARV Agent (Cohort 1) (N=28) | F/TAF+3rd ARV Agent (Cohort 2, Part A - Group 1) (N=9) | F/TAF+3rd ARV Agent (Cohort 2, Part A - Group 2) (N=3)
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 4 | 2 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1
Eczema eyelids (Eye disorders) | 0 | 1 | 0
Vernal keratoconjunctivitis (Eye disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 3 | 0 | 0
Dental caries (Gastrointestinal disorders) | 4 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 6 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 3 | 0 | 0
Nausea (Gastrointestinal disorders) | 6 | 0 | 0
Vomiting (Gastrointestinal disorders) | 7 | 1 | 0
Pyrexia (General disorders) | 2 | 0 | 0
Acarodermatitis (Infections and infestations) | 2 | 0 | 0
Bacterial vaginosis (Infections and infestations) | 2 | 0 | 0
Body tinea (Infections and infestations) | 4 | 0 | 0
Conjunctivitis (Infections and infestations) | 3 | 0 | 0
Covid-19 (Infections and infestations) | 2 | 2 | 0
Folliculitis (Infections and infestations) | 2 | 0 | 0
Gastroenteritis (Infections and infestations) | 4 | 2 | 0
Gastroenteritis viral (Infections and infestations) | 2 | 0 | 0
Helminthic infection (Infections and infestations) | 0 | 0 | 1
Hordeolum (Infections and infestations) | 3 | 1 | 0
Influenza (Infections and infestations) | 8 | 1 | 0
Nasopharyngitis (Infections and infestations) | 13 | 5 | 0
Otitis externa (Infections and infestations) | 1 | 1 | 0
Otitis media acute (Infections and infestations) | 2 | 0 | 0
Pharyngitis (Infections and infestations) | 5 | 1 | 1
Pharyngotonsillitis (Infections and infestations) | 0 | 2 | 0
Pneumonia (Infections and infestations) | 2 | 0 | 0
Respiratory tract infection (Infections and infestations) | 3 | 0 | 0
Sinusitis (Infections and infestations) | 2 | 0 | 0
Tonsillitis (Infections and infestations) | 2 | 0 | 0
Tooth abscess (Infections and infestations) | 3 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 7 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 2 | 0 | 2
Vulvovaginal mycotic infection (Infections and infestations) | 2 | 0 | 0
Animal bite (Injury, poisoning and procedural complications) | 2 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 3 | 0 | 0
Heat stroke (Injury, poisoning and procedural complications) | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 2 | 0 | 0
Seroma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 1 | 0
Vitamin D decreased (Investigations) | 0 | 1 | 0
Weight decreased (Investigations) | 5 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 7 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Dizziness (Nervous system disorders) | 6 | 0 | 0
Headache (Nervous system disorders) | 13 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 1
Adjustment disorder (Psychiatric disorders) | 2 | 0 | 0
Depression (Psychiatric disorders) | 5 | 0 | 0
Insomnia (Psychiatric disorders) | 3 | 0 | 0
Haematuria (Renal and urinary disorders) | 2 | 0 | 0
Balanoposthitis (Reproductive system and breast disorders) | 1 | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 2 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 2 | 0 | 0
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Respiratory symptom (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 0
Acne (Skin and subcutaneous tissue disorders) | 8 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Circumcision (Surgical and medical procedures) | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (3):
  • Study Protocol (2017-08-02): https://cdn.clinicaltrials.gov/large-docs/14/NCT02285114/Prot_002.pdf
  • Statistical Analysis Plan: Interim Analysis (2020-10-06): https://cdn.clinicaltrials.gov/large-docs/14/NCT02285114/SAP_001.pdf
  • Statistical Analysis Plan: Final Analysis (2025-02-19): https://cdn.clinicaltrials.gov/large-docs/14/NCT02285114/SAP_003.pdf